CLINICAL TRIAL: NCT04450017
Title: Clinical Features of Severe Patients With COVID-19
Status: Completed | Type: Observational
Sponsor: Federal Research Clinical Center of Federal Medical & Biological Agency, Russia (Other Government)
Responsible Party: Sponsor
Other Study IDs: COVID-ICU
Record Dates: First submitted 2020-06-23; First posted 2020-06-29 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: SARS-CoV2
Keywords: SARS pneumonia; COVID-19; severe disease; risk factors
MeSH Terms: conditions — COVID-19; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Clinical Features of Severe Patients With COVID-19: Critical ill patients with COVID-19 admitted to the ICU. The demographic, clinical data, laboratory data, and Instrumental data will be analysed.
  Interventions: Diagnostic Test: The demographic, clinical, laboratory, and instrumental data

INTERVENTIONS:
Diagnostic Test: The demographic, clinical, laboratory, and instrumental data — Measurement of the demographic, clinical data, laboratory data, and instrumental data

SUMMARY:
As coronavirus disease 2019 (COVID-19) spreads across the world, the intensive care unit (ICU) community must prepare for the challenges associated with this pandemic. Providing an efficient care to the patients of the most severely affected category - intensive care unit (ICU) patients - has become one of the serious problems appearing in the COVID-19 pandemics. A typical patient's clinical portrait in ICU of COVID centers is very similar in different countries, however, the key to improve the treatment results for critically ill patients has not yet been found. Data on predictors of severe course in COVID-19 is limited. Knowledge of predictors of severe course of disease can lead to different selection of therapeutic strategy, determine the group of risk of patients for severe course of disease, and improve outcomes.

DETAILED DESCRIPTION:
The clinical disease (COVID-19) results in critical illness in about 5% of patients. The aim of the study is to identify predictors of the severe pneumonia caused by the SARS-CoV-2 virus, and to describe the clinical features of patients admitted to an ICU of the COVID-center of the Federal Research Clinical Center of Federal Medical & Biological Agency on the first day and in dynamics till discharge from the ICU or death.

The demographic and clinical data will be collected. Laboratory data (hemoglobin, lymphocytes, neutrophil to lymphocyte ratio, D-dimer level, IL-6, procalcitonin, glucose level, high-sensitive troponin Т, vitamin D level, signs of the presence of a secondary bacterial infection, immunogram and Instrumental data (CT-scan, Electrocardiography, echocardiography, arterial and venous ultrasound investigation) will be analysed.

This study is singlecentral observational trial.

ELIGIBILITY:
Inclusion Criteria:

* all patients with COVID-19 admitted to the ICU with invasive and noninvasive ventilation

Exclusion Criteria:

* less than 24 hours in ICU by any reason,
* chronic decompensated diseases with extrapulmonary organ dysfunction (tumour progression, liver cirrhosis, congestive heart failure),
* atonic coma.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with COVID-19 requiring respiratory support
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-04-06 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Mechanical ventilation duration | 30 days
  The amount of mechanical ventilation days
Non-invasive Mechanical ventilation duration | 30 days
  The amount of Non-invasive mechanical ventilation days
Mortality | 60 days
  The dead and survived patients ratio

SECONDARY OUTCOMES:
Сomplete blood count | Change from baseline on day 5 during ICU treatment
  Сomplete blood count
Biochemistry analysis | Change from baseline on day 5 during ICU treatment
  Biochemistry analysis
Сomplete blood count dynamics | Change from baseline on day 15 during ICU treatment
  Сomplete blood count
Biochemistry analysis dynamics | Change from baseline on day 15 during ICU treatment
  Biochemistry analysis
Computer tomography | Change from baseline on day 5 during ICU treatment
  Computer tomography of lungs
High-sensitive troponin Т | Change from baseline on day 5 during ICU treatment
  High-sensitive troponin Т
High-sensitive troponin Т dynamics | Change from baseline on day 15 during ICU treatment
  High-sensitive troponin Т
Vitamin D level | Change from baseline on day 5 during ICU treatment
  Vitamin D level
Vitamin D level dynamics | Change from baseline on day 15 during ICU treatment
  Vitamin D level
Immunogram | Change from baseline on day 5 during ICU treatment
  Immunogram
Immunogram dynamics | Change from baseline on day 15 during ICU treatment
  Immunogram

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana V Klypa, Dr.Med.Sc., Principal Investigator — Federal Research Clinical Center of Federal Medical & Biological Agency
Locations (1):
- Federal Research Clinical Center of Federal Medical & Biological Agency, Moscow, Russia

REFERENCES:
- [Background] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Background] Tian W, Jiang W, Yao J, Nicholson CJ, Li RH, Sigurslid HH, Wooster L, Rotter JI, Guo X, Malhotra R. Predictors of mortality in hospitalized COVID-19 patients: A systematic review and meta-analysis. J Med Virol. 2020 Oct;92(10):1875-1883. doi: 10.1002/jmv.26050. Epub 2020 Jul 11. PMID 32441789
- [Background] Paranjpe I, Russak AJ, De Freitas JK, Lala A, Miotto R, Vaid A, Johnson KW, Danieletto M, Golden E, Meyer D, Singh M, Somani S, Manna S, Nangia U, Kapoor A, O'Hagan R, O'Reilly PF, Huckins LM, Glowe P, Kia A, Timsina P, Freeman RM, Levin MA, Jhang J, Firpo A, Kovatch P, Finkelstein J, Aberg JA, Bagiella E, Horowitz CR, Murphy B, Fayad ZA, Narula J, Nestler EJ, Fuster V, Cordon-Cardo C, Charney DS, Reich DL, Just AC, Bottinger EP, Charney AW, Glicksberg BS, Nadkarni GN. Clinical Characteristics of Hospitalized Covid-19 Patients in New York City. medRxiv [Preprint]. 2020 Apr 26:2020.04.19.20062117. doi: 10.1101/2020.04.19.20062117. PMID 32511655
- [Derived] Bychinin MV, Klypa TV, Mandel IA, Andreichenko SA, Baklaushev VP, Yusubalieva GM, Kolyshkina NA, Troitsky AV. Low Circulating Vitamin D in Intensive Care Unit-Admitted COVID-19 Patients as a Predictor of Negative Outcomes. J Nutr. 2021 Aug 7;151(8):2199-2205. doi: 10.1093/jn/nxab107. PMID 33982128